CLINICAL TRIAL: NCT05716243
Title: Effect of Nociception Level Index on Postoperative Pain Management in Pediatric Patients
Brief Title: Nociception Level Index as a Verbal Tool of Pain in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 211-2022
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Pediatric Patients; Orthopedic Surgery; Extremity Fractures Lower; Extremity Fractures Upper; Deformity; Congenital
Keywords: postoperative pain; nociception level index; behavioral pain scores; general anesthesia; pain monitorization
MeSH Terms: conditions — Congenital Abnormalities; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: After standard monitorization, general anesthesia will be applied. Once the randomization is concluded to decide the group of the patient, Group A will receive 15 mg/kg (IV) paracetamol and 0,05 mg/kg morphine (IV). For once, NOL monitorization will be applied 30 minutes before waking up the patient to assess standard pain management and if the NOL value is higher than 25; 0,025 mg/kg morphine (IV) bolus doses (the maximum total intraoperative dose is concluded to be 0,5 mg/kg (IV)) will be added to ensure adequate analgesia for all patients within the study. On the contrary, patients within Group B will receive NOL monitorization from the beginning, all along the surgery.
Who Masked: Outcomes Assessor
Masking Description: The anesthetist who is blind to study groups will make all postoperative assessments of pain by FLACC (Face, Legs, Activity, Cry, Consolability) behavioral pain assessment score at the postoperative care unit, 6th 12th, and 24th hour postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A will receive a standard intraoperative analgesia protocol
  Interventions: Device: The nociception level index measurement;postoperative
- Group B (Experimental): Group B will receive a NOL-guided analgesia protocol
  Interventions: Device: The nociception level index monitorization

INTERVENTIONS:
Device: The nociception level index monitorization — The nociception level index (NOL) is one of the nociception monitors and stands out from the others with its multi-parameter evaluation. It is generated from five different parameters (heart rate, heart rate variability, skin conductance level, photo-plethysmography waveform amplitude, number of skin conductance fluctuations, and their time derivatives).
  Arms: Group B
Device: The nociception level index measurement;postoperative — The nociception level index (NOL) will be used postoperatively
  Arms: Group A

SUMMARY:
60 children under 6 years old, scheduled for orthopedic surgery for limb fracture or neuromuscular and bone deformities will be randomized by closed envelope method into two groups (n=30) either receiving standard pain management protocol or intraoperative NOL guided analgesia. Our study aims to evaluate the nociception monitor's effectiveness in providing adequate postoperative analgesia in pediatric patients. Besides, the difference between the amount of analgesic medication will be recorded.

Data to be recorded are total intraoperative morphine and postoperative rescue analgesic consumption, NOL values, and FLACC scores.

DETAILED DESCRIPTION:
The nociception level index (NOL) is one of the nociception monitors and stands out from the others with its multi-parameter evaluation. It is generated from five different parameters (heart rate, heart rate variability, skin conductance level, photo-plethysmography waveform amplitude, number of skin conductance fluctuations, and their time derivatives). Moreover, its design as a finger probe connected to a non-invasive continuous nociception monitor makes it more suitable, especially for pediatric patients. Although this monitor has been validated for discrimination of a noxious stimulus with high accuracy, its effects on perioperative pain management have recently started to be shown in clinical practice. More importantly, no study has yet been conducted on the use of NOL monitoring in pain management in pediatric patients.

The study is designed as a single-blind, prospective study after approval of our Institutional ethics committee (dossier no:211-2022) and planned to allocate 60 patients (2 groups; 1:1 allocation; n=30) after obtaining written informed parental consent. Children aged under 6 who are scheduled for orthopedic surgery for limb fracture or neuromuscular and bone deformities are eligible for this study. Exclusion criteria are refusal to participate in the study; history of premature birth; known metabolic syndrome; allergies to drugs used within the study protocol; decreased liver or renal function; diagnosed mental retardation.

Patient randomization Randomization is designed with concealed opaque envelope in a 1:1 ratio into 2 groups (n= 30): the control group (Group A) and the study group (Group B). Before the start of the study, an independent anesthetist will prepare 60 envelopes each containing the name of one group. When the inclusion/exclusion criteria are met, on the day of the surgery the anesthetist will choose one envelope in the operating room to apply the designed protocol for each group. Data obtained at the clinical follow-up will be gathered by an independent anesthetist who is blinded to the groups and protocol used in the operating room.

Anesthesia, intervention, and post-interventional follow-up After standard monitorization, general anesthesia induction will start with sevoflurane 4-6% administered via a face mask. Subsequently, after intravenous (IV) cannulation 2 mcg/kg fentanyl; 0,05 mg/kg midazolam; 1-2,5 mg/kg propofol; 0,6 mg/kg rocuronium will be administered and orotracheal intubation will be performed. Once the randomization is concluded to decide the group of the patient, Group A will receive 15 mg/kg (IV) paracetamol and 0,05 mg/kg morphine (IV). For once, NOL monitorization will be applied 30 minutes before waking up the patient to assess standard pain management and if the NOL value is higher than 25; 0,025 mg/kg morphine (IV) bolus doses (the maximum total intraoperative dose is concluded to be 0,5 mg/kg (IV)) will be added to ensure adequate analgesia for all patients within the study. On the contrary, patients within Group B will receive NOL monitorization from the beginning, all along the surgery. As pain management protocol, other than standard 15 mg/kg (IV) paracetamol, 0,025 mg/kg morphine (IV) bolus doses will be applied if only intraoperative NOL values are over 25 (concluded to be valuable only if it remains over 25 for at least one minute). Postoperative pain was assessed by FLACC (Face, Legs, Activity, Cry, Consolability) behavioral pain assessment score at the postoperative care unit, 6th 12th, and 24th hour postoperatively. The same anesthetist who is blind to study groups will make all assessments to precise standardization. All children will be prescribed paracetamol 15 mg/kg (IV) four times per day. If the pain score was equal to or more than 4, tramadol 1 mg/kg will be administered intravenously as a rescue analgesic. The amount of total intraoperative morphine and postoperative rescue analgesic consumption along with NOL values and FLACC scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) Physical Status classification I to II
* Patients whose parents will give informed consent for the study

Exclusion Criteria:

* Refusal to take part in the study
* History of allergies to drugs used in the study protocol
* History of premature birth
* Diagnosed metabolic syndrome
* Known hepatic insufficiency or decreased function
* Known renal insufficiency or decreased function
* Diagnosed with mental retardation

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Pain Scores | postoperative 24 hour
  Face, Legs, Activity, Cry, Consolability (FLACC) behavioral pain assessment score : range 0-10; 0 = Relaxed and comfortable;1-3 = Mild discomfort; 4-6 = Moderate. pain.
  7-10 = Severe discomfort/pain.

SECONDARY OUTCOMES:
The total amount of analgesic drug | Intraoperative and postoperative 24 hour
  morphine(mg) used intraoperatively and tramadol(mg) at postoperative follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, MD, Principal Investigator — Haseki Training and Research Hospital Anesthesiology and Reanimation Department
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gomez-Rios MA, Abad-Gurumeta A, Calvo-Vecino JM. Assessing nociception: steps towards intraoperative "full monitoring". Minerva Anestesiol. 2018 Oct;84(10):1123-1125. doi: 10.23736/S0375-9393.18.13191-9. No abstract available. PMID 30274508
- [Result] Ghiyasinasab M, Morisson L, Laferriere-Langlois P, Geraldo-Demers MA, Gelinas C, Nadeau-Vallee M, Verdonck O, Lahrichi N, Richebe P. Identification of the intraoperative antinociceptive effect of intravenous fentanyl using the Nociception Level (NOL) index versus clinical parameters in patients undergoing gynecological laparoscopic surgery: A secondary analysis of the NOLGYN study. Anaesth Crit Care Pain Med. 2022 Aug;41(4):101102. doi: 10.1016/j.accpm.2022.101102. Epub 2022 May 25. PMID 35643392
- See also: Assessment of Pain in Children Shobha Malviya MD University of Michiga — https://www2.pedsanesthesia.org/meetings/2006annual/syllabus/AssessmentofPain-Malviya.pdf